CLINICAL TRIAL: NCT03728530
Title: Effect Of Deep Breathing Exercises In Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isra University (Other)
Responsible Party: Principal Investigator, Noor Abid, Research Associate, Isra University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIRS-IUISB/DPT/024
Record Dates: First submitted 2018-01-11; First posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-11

CONDITIONS: Healthy Smokers
Keywords: Deep breathing exercises, smokers, lung function

STUDY DESIGN:
Intervention Model Description: Study was to determine the effects of deep breathing exercises in smokers. It was conducted on the general population of Isra Institute of Rehabilitation Sciences, Isra University, Islamabad Campus. 30 participants were selected through Non probability Convenience Sampling and later equally divided into experimental (n=15) and control group (n=15) through lottery method. Inclusion criteria were young smokers between 20-30 years of age and without any chronic pulmonary complication, smoking for past five years. Smokers with any pulmonary disease, acute infections, other systemic disease, chest deformity or any disability were excluded from study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Deep /breathing exercises including Purse lip, diaphragmatic breathing and powered breathing
  Interventions: Other: Deep Breathing exercises
- Control Group (No Intervention): The participants from control group did not perform any exercise.

INTERVENTIONS:
Other: Deep Breathing exercises — In pursed lip exercise subject was guided to inhale through nose with mouth closed and exhale through pressed lips (pursed lips).
  In Diaphragmatic breathing subject was instructed to place his one hand below the rib cage and the other hand on chest. The patient inhaled slowly so that stomach moves out against the hand. Tighten the stomach muscle while exhaling through pursed lip.
  In powered breathing subject was to inhale and exhale forcefully with some movements like subject was instructed to inhale forcefully while moving his hands upward and exhale forcefully while moving hands downward.
  These three exercise techniques were advised to each subject of experimental group. They have to practice these exercises 3-4 times a day with 10 repetitions each. These exercises can be performed in sitting position or in supine lying position. Subject can adopt any position in which he feels comfortable.
  Arms: Experimental Group

SUMMARY:
To determine the effect of deep breathing exercises on lung function in healthy smokers.

DETAILED DESCRIPTION:
The purpose of the study to determine the effect of deep breathing exercise in smokers because deep breathing improve the lung capacity by filling the lung with the oxygen and improve the pulmonary function, it also reduce the stress and anxiety level by slowing down the pace of your whole body and therefore promote general relaxation and improve the quality of life in smokers, muscular activity or physical activity is also increased because by deep breathing maximum oxygen is reached to every muscle and they get nourish well so overall impact of deep breathing exercise is positive. Deep breathing exercise technique offered in the study are easy to learn and can be performed by everyone and everywhere safely, because there is no complex and pain full procedure. So deep breathing exercise have been proposed as a way of combating cigarette craving, improves quality of life and lung function.

ELIGIBILITY:
Inclusion Criteria:

Young male and female adults with age group of 20-30 years without any chronic complication doing smoking from past five years are included in this study as the basic purpose of the study is to determine the effects of deep breathing exercises in smokers

Exclusion Criteria:

1. Adults with pulmonary disease.
2. Acute infections
3. Any other systemic disease.
4. Chest deformity.
5. Adults with any disability.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2017-02-22 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Oxygen Saturation | 2 weeks
  Pulse Oximetry was used to measure oxygen saturation
Lung Volumes | 2 weeks
  All lung volume were measured with spirometer
Lung Capacities | 2 weeks
  All lung capacities were measured with spirometer

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available within a month